CLINICAL TRIAL: NCT05987085
Title: Effect of Medical Weight Loss on Pelvic Floor Dysfunction: a Prospective Observational Study
Brief Title: Medical Weight Loss on Pelvic Floor Dysfunction
Acronym: WLPFD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhijing Sun, Professor, Peking Union Medical College Hospital
Other Study IDs: WLPFD-PUMCH
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-08

CONDITIONS: Weight Loss; Pelvic Floor Disorders
MeSH Terms: conditions — Weight Loss; Pelvic Floor Disorders | interventions — Diet; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diet and exercise — Routine intervention included diet control and exercise

SUMMARY:
The goal of this observational study is to learn about the effect of medical weight loss on the symptom of pelvic floor dysfunction in obese and overweight women. The main question it aims to answer is: whether medical weight loss improves symptoms of pelvic floor dysfunctions in obese or overweight women.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or higher
* BMI 24 kg/m2 or higher
* Willing to follow the weight loss plan set by the physician follow-up and complete this study

Exclusion Criteria:

* Urinary tract infection or gynecologic reproductive system infection in the past month
* Treatment history of pelvic floor disorders
* Pregnancy or delivery in the past half year
* Women with severe systemic disease
* No follow-up conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women seeking medical weight loss
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor symptoms before and after medical weight loss | At least half a year

SECONDARY OUTCOMES:
To explore the related factors of symptom improvement in pelvic floor dysfunction | At least half a year
To explore the improvement of quality of life before and after medical weight loss | At least half a year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Z, Chen W, Sun Z. Protocol for a prospective longitudinal cohort study on the effects of non-surgical weight loss on pelvic floor dysfunction. BMJ Open. 2024 Feb 5;14(2):e079143. doi: 10.1136/bmjopen-2023-079143. PMID 38316600